CLINICAL TRIAL: NCT04111679
Title: The Effect of Preferred Music on Laparoscopic Performance
Brief Title: EffectS of prEferred Music on Laparoscopic performancE
Acronym: EnSEMbLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. dr. Gert-Jan Kleinrensink, Professor of anatomy, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC-2018-1134
Record Dates: First submitted 2019-09-04; First posted 2019-10-01 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Laparoscopic Surgery; Music; Surgical Education
Keywords: Surgical skill; Music; Laparoscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: This will be a 4-period 4-sequence 2-treatment crossover study, participants will be exposed to both control group (A), the silent group, and intervention group (B), the music group, whilst performing a laparoscopic task in a box trainer.
  Participants will be randomly assigned to a sequence that determines in which order they are being exposed to both auditory environments
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): During laparoscopic task performance; participants will wear a noise cancelling headphone that plays music that is chosen by the participant.
  Interventions: Other: Music
- No music (No Intervention): During laparoscopic task performance; participants will wear a noise cancelling headphone that does not play music.

INTERVENTIONS:
Other: Music — Participant selected music, applied using noise cancelling headphones
  Arms: Music

SUMMARY:
The main objective is to investigate whether listening to recorded music has a positive effect on the execution of laparoscopic skills.

Secondary objectives are to investigate the effects of music during surgical performance on blood pressure, mental workload and heart rate.

Study design: This will be a 4-period 4-sequence 2-treatment crossover study, participants will be exposed to both control (noise cancelling headphones without music) and the intervention (preferred music via headphones) whilst performing a laparoscopic task in a box trainer. Every period consists of 5 repetitions of a laparoscopic peg transfer task. In total participants will perform in each condition 10 peg transfer tasks.

Prior to the experiment, all participants practice the laparoscopic peg transfer task 20 times

Study population: Healthy volunteering medicine students without laparoscopic experience.

Intervention (if applicable): Participants will perform 2 periods of 5 laparoscopic peg transfer task whilst listening to preferred recorded music via headphones and 2 periods of 5 laparoscopic peg transfer tasks while wearing noise cancelling headphones without music (2 periods of 5 tasks).

Main study parameters/endpoints: The primary endpoint is laparoscopic performance as defined by time of task completion Secondary endpoints are: laparoscopic task performance (path length, jerk, error score, economy of motion) vital parameters (heart rate, and post test blood pressure) and mental workload (SURG-TLX)

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study a subject must meet all of the following criteria.

* Age ≥ 18 years
* Medicine students
* Provision of written informed consent by the subject.

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Severe hearing impairment, defined as no verbal communication possible.
* Severe visual impairment, defined as not able to see the monitor on which the laparoscopic task is projected.
* Any physical handicap that impairs laparoscopic performance (unable to stand for 10 minutes, unable to hold and use both instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Time to task completion (s) | This will be measured during the experimental session which will take up about 1 hour in total
  It will be measured in seconds and calculated using data generated from motion analysis software. Each tasks starts, when the participants puts the tip of the grasper in a yellow square that is projected on the screen, after task completion the participant puts tip in the square again to finish the task. The time between start and finish is defined as the time to task completion.
  An average is calculated for both the 10 tasks in the intervention group and the 10 tasks in the control group.

SECONDARY OUTCOMES:
Path length | This will be measured during the experimental session which will take up about 1 hour in total
  The total distance the tip of the instrument has travelled per task (mm) per task, it will be calculated using data generated from motion analysis software. Each tasks starts, when the participants puts the tip of the grasper in a yellow square that is projected on the screen, after task completion the participant puts tip in the square again to finish the task. An average is calculated for both the 10 tasks in the intervention group and the 10 tasks in the control group.
Normalized jerk | This will be measured during the experimental session which will take up about 1 hour in total
  the rate of change of acceleration of the instrument tips (m/s3) per task. It will be calculated using data generated from motion analysis software. Each tasks starts, when the participants puts the tip of the grasper in a yellow square that is projected on the screen, after task completion the participant puts tip in the square again to finish the task. An average is calculated for both the 10 tasks in the intervention group and the 10 tasks in the control group.
Mental workload | This will be measured during the experimental session which will take up about 1 hour in total
  Mental workload will be assessed using the Surgery task load index (SURG-TLX) this is a validated multidimensional, surgery-specific workload measure. The SURG-TLX is an adapted version of the National Aeronautics and Space Administration Task Load Index (NASA-TLX).
  In the SURG-TLX subjects rate six dimensions of workload i.e. situational stress, distractions, task complexity, physical demands, temporal demands and mental demands on visual analogue scales VAS ranging from 0-100 (0 = very low;100 = very high) the scores of these subscales are combined into a weighed average that results in a general score ranging from 0-100 (0 = very low; 100 = very high) After every period of 5 tasks a SURG-TLX questionnaire is completed. An average is calculated for both the two periods in the intervention group and the two periods in the control group. The averages of both the general score and the individual subscales will be reported.
Heart rate | This will be measured during the experimental session which will take up about 1 hour in total
  Heart rate will be assessed prior to; and immediately after every period of laparoscopic tasks in beats per minute. Change in heart rate before and after each period of tasks is calculated. An average change will be calculated for both the two periods in the intervention group and the two periods in the control group
Blood pressure | This will be measured during the experimental session which will take up about 1 hour in total
  Systolic and diastolic pressure will be assessed prior to and immediately after every period of laparoscopic tasks in mmHg. Change in blood pressure before and after each period of tasks is calculated. An average change will be calculated for both the two periods in the intervention group and the two periods in the control group
Participant's characteristics | This will be measured during the experimental session which will take up about 1 hour in total
  * Age (years)
  * Sex (male or female)
  * Dexterity (left- or right handed, ambidextrous)
  * Year of medical education:
  * The importance of music in daily life on a (10-point numeric rating scale)
  * Musical genres the subject listens to (classical, world music, rock, pop, techno, house, jazz, blues, disco, other)
  * Musical genres the subject listens to when studying: (classical, world music, rock, pop, techno, house, jazz, blues, disco, other)
  * choice of music during the experiment
  * Whether or not the subject plays or has played a musical instrument (never, in the past, currently)
  * Whether or not the subject plays or has played video games and to what extends (never, in the past, currently)
  This questionnaire will be completed before starting the practice session of 20 laparoscopic tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Gert-Jan Kleinrensink, Prof. Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oomens P, Fu VX, Kleinrensink VEE, Kleinrensink GJ, Jeekel J. The Effects of Preferred Music on Laparoscopic Surgical Performance: A Randomized Crossover Study. World J Surg. 2020 Aug;44(8):2614-2619. doi: 10.1007/s00268-020-05523-0. PMID 32333159